CLINICAL TRIAL: NCT03519971
Title: A Phase III, Randomized, Placebo-controlled, Double-blind, Multi-center, International Study of Durvalumab Given Concurrently With Platinum-based Chemoradiation Therapy in Patients With Locally Advanced, Unresectable NSCLC (Stage III) (PACIFIC2)
Brief Title: Study of Durvalumab Given With Chemoradiation Therapy in Patients With Unresectable Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D933KC00001; 2017-004397-34 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-05-09 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally Advanced, Unresectable NSCLC, Carcinoma, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — durvalumab; PE regimen; CP protocol; Pemetrexed; Cisplatin; Carboplatin; Radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Durvalumab + platinum-based chemotherapy and radiation (Experimental): Durvalumab ((MEDI4736) in concurrence with platinum-based chemo-radiation therapy.
  All patients will receive 1 of the following platinum-based standard of care chemotherapy options, based on Investigator discretion, in addition to radiation therapy:
  * cisplatin/etoposide
  * carboplatin/paclitaxel
  * pemetrexed/cisplatin
  * pemetrexed/carboplatin
  At the completion of standard of care chemoradiation therapy (SoC CRT), patients with complete response, partial response or stable disease will continue to receive durvalumab as consolidation treatment.
  Interventions: Drug: Durvalumab; Drug: Cisplatin/ Etoposide; Drug: Carboplatin/ Paclitaxel; Drug: Pemetrexed/ Cisplatin; Drug: Pemetrexed/ Carboplatin; Radiation: Radiation
- Arm 2: Placebo + platinum-based chemotherapy and radiation (Placebo Comparator): Placebo in concurrence with platinum-based chemo-radiation therapy.
  All patients will receive 1 of the following platinum-based standard of care chemotherapy options, based on Investigator discretion, in addition to radiation therapy:
  * cisplatin/etoposide
  * carboplatin/paclitaxel
  * pemetrexed/cisplatin
  * pemetrexed/carboplatin
  At the completion of standard of care chemoradiation therapy (SoC CRT), patients with complete response, partial response or stable disease will continue to receive placebo as consolidation treatment.
  Interventions: Other: Placebo; Drug: Cisplatin/ Etoposide; Drug: Carboplatin/ Paclitaxel; Drug: Pemetrexed/ Cisplatin; Drug: Pemetrexed/ Carboplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion)
  Other Names: MEDI4736
  Arms: Arm 1: Durvalumab + platinum-based chemotherapy and radiation
Other: Placebo — Placebo IV (intravenous infusion)
  Arms: Arm 2: Placebo + platinum-based chemotherapy and radiation
Drug: Cisplatin/ Etoposide — Cisplatin/ Etoposide, as per standard of care
Drug: Carboplatin/ Paclitaxel — Carboplatin /Paclitaxel, as per standard of care
Drug: Pemetrexed/ Cisplatin — Pemetrexed / Cisplatin, as per standard of care
Drug: Pemetrexed/ Carboplatin — Pemetrexed / Carboplatin , as per standard of care
Radiation: Radiation — 5 fractions/ week for ~6 weeks (±3 days) (Total 60 Gy)

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled, multi-center, international study assessing the efficacy and safety of durvalumab given concurrently with platinum-based CRT (durvalumab + standard of care [SoC] CRT) in patients with locally advanced, unresectable NSCLC (Stage III).

ELIGIBILITY:
Principal inclusion criteria :

* Subjects with histologically- or cytologically-documented NSCLC
* Locally advanced, unresectable (Stage III) NSCLC
* World Health Organisation (WHO) performance status 0-1
* At least one measurable lesion, not previously irradiated
* Must have a life expectancy of at least 12 weeks at randomization

Principal exclusion criteria :

* Receipt of prior or current cancer treatment, including but not limited to, radiation therapy, investigational agents, chemotherapy, Durvalumab and mAbs.
* Prior exposure to immune-mediated therapy, including but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti PD L2 antibodies, excluding therapeutic anticancer vaccines.
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders
* Uncontrolled intercurrent illness
* History of another primary malignancy / leptomeningeal carcinomatosis / active primary immunodeficiency
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus
* Mixed small cell and NSCLC histology
* Any medical contraindication to treatment with platinum-based doublet chemotherapy as listed in the local labelling
* Known allergy or hypersensitivity to any of the IPs or any of the IP excipients.
* Patients whose radiation treatment plans are likely to encompass a volume of whole lung receiving ≥20 Gy in total (V20) of more than 35% of lung volume.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2025-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, MD, Principal Investigator — AstraZeneca
Locations (71):
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Czechia (3):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Prague
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Törökbálint
- India (8):
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Gūrgaon
  - Research Site, Karamsad
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Vadodara
- Japan (8):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Nagoya
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Yokohama
- Mexico (6):
  - Research Site, Aguascalientes
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Orizaba
- Peru (2):
  - Research Site, La Libertad
  - Research Site, Lima
- Philippines (6):
  - Research Site, Cebu City
  - Research Site, City of Taguig
  - Research Site, Iloilo City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Olsztyn
  - Research Site, Warsaw
- Russia (6):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
- South Korea (4):
  - Research Site, Busan
  - Research Site, Chungcheongbuk-do
  - Research Site, Gyeongsangnam-do
  - Research Site, Seoul
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Mueang
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Diyarbakır
  - Research Site, Istanbul
  - Research Site, Izmir
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933KC00001&attachmentIdentifier=c84b8a9a-ab3b-42d9-beef-8e42857afd0d&fileName=D933KC00001_-___Statistical_Analysis_Plan_-_Redacted.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933KC00001&attachmentIdentifier=734b41e6-780c-402f-a50f-4a03f71afabb&fileName=D933KC00001_-_Protocol_-_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933KC00001&attachmentIdentifier=ed59b3e6-e0a6-4b8b-96e1-49b8ff510ee7&fileName=D933KC00001_-_Study_Synopsis_-_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III double-blind, placebo-controlled study was conducted in participants with locally advanced, unresectable Stage III non-small cell lung cancer (NSCLC) at 87 study centers in North and South America, Europe, and Asia Pacific. The results are reported for analysis with assessment until data cut-off (DCO) date of 07 September 2023.
Pre-assignment Details: The study had a screening period (up to 28 days), followed by a treatment and follow-up period (up to 1960 days). A total of 328 participants were randomized in a 2:1 ratio to receive durvalumab + standard of care (SoC) concurrent chemoradiotherapy (cCRT) group or placebo + SoC cCRT group.
Groups:
- Durvalumab + SoC CRT: Participants received durvalumab 1500 milligram (mg) intravenous (IV) infusion every 4 weeks (Q4W) until progressive disease (PD) or specific treatment discontinuation criteria were met.
  Participants received SOC CRT, consisting of concurrent radiotherapy and IV infusion of 1 of the following chemotherapy regimens.
  1. Cisplatin + Etoposide: Cisplatin 50 mg/square meter (m^2) on Days 1 and 8 and etoposide 50 mg/m^2 on Days 1 to 5 Q4W of each 28-day cycle for 2 cycles plus 1 additional optional induction cycle.
  2. Carboplatin + Paclitaxel: Carboplatin area under the plasma drug concentration-time curve (AUC) 2 and paclitaxel 40-50 mg/m^2 on Day 1 weekly basis for 6 weeks. Optional: Carboplatin AUC 5-6 and paclitaxel 175-200 mg/m^2 every 3 weeks (Q3W) given either as 1 induction cycle prior to initiation of radiation therapy (RT) or as 1-2 consolidation cycles after completion of RT.
  3. Cisplatin + Pemetrexed: Cisplatin 75 mg/m^2 and pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for 3 cycles plus 1 additional optional induction cycle.
  4. Carboplatin + Pemetrexed: Carboplatin AUC 5 and pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for 4 cycles.
  Radiation: Either standard 3-dimensional conformal radiotherapy (3DCRT) or intensity-modulated radiation therapy (IMRT) was delivered using external beam radiation therapy (EBRT) of 5 fractions per week for ~6 weeks (± 3 days).
- Placebo + SoC CRT: Participants received placebo matching with durvalumab IV infusion Q4W until PD or specific treatment discontinuation criteria were met.
  Participants received SOC CRT, consisting of concurrent radiotherapy and IV infusion of 1 of the following chemotherapy regimens.
  1. Cisplatin + Etoposide: Cisplatin 50 mg/m^2 on Days 1 and 8 and etoposide 50 mg/m^2 on Days 1 to 5 Q4W of each 28-day cycle for 2 cycles plus 1 additional optional induction cycle.
  2. Carboplatin + Paclitaxel: Carboplatin AUC 2 and paclitaxel 40-50 mg/m^2 on Day 1 weekly basis for 6 weeks. Optional: Carboplatin AUC 5-6 and paclitaxel 175-200 mg/m^2 Q3W given either as 1 induction cycle prior to initiation of RT or as 1-2 consolidation cycles after completion of RT.
  3. Cisplatin + Pemetrexed: Cisplatin 75 mg/m^2 and pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for 3 cycles plus 1 additional optional induction cycle.
  4. Carboplatin + Pemetrexed: Carboplatin AUC 5 and pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for 4 cycles.
  Radiation: Either standard 3DCRT or IMRT was delivered using EBRT of 5 fractions per week for ~6 weeks (± 3 days).
Period: Overall Study
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Started | 219 | 109
Received Treatment | 218 | 109
Completed | 0 | 0
Not Completed | 219 | 109
Not completed — Death | 142 | 69
Not completed — Lost to Follow-up | 0 | 1
Not completed — Ongoing treatment and in follow-up at data cut off | 73 | 37
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomized participants.
Groups:
- Durvalumab + SoC CRT: Participants received durvalumab 1500 mg IV infusion Q4W until PD or specific treatment discontinuation criteria were met.
  Participants received SOC CRT, consisting of concurrent radiotherapy and IV infusion of 1 of the following chemotherapy regimens.
  1. Cisplatin + Etoposide: Cisplatin 50 mg/m^2 on Days 1 and 8 and etoposide 50 mg/m^2 on Days 1 to 5 Q4W of each 28-day cycle for 2 cycles plus 1 additional optional induction cycle.
  2. Carboplatin + Paclitaxel: Carboplatin AUC 2 and paclitaxel 40-50 mg/m^2 on Day 1 weekly basis for 6 weeks. Optional: Carboplatin AUC 5-6 and paclitaxel 175-200 mg/m^2 Q3W given either as 1 induction cycle prior to initiation of RT or as 1-2 consolidation cycles after completion of RT.
  3. Cisplatin + Pemetrexed: Cisplatin 75 mg/m^2 and pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for 3 cycles plus 1 additional optional induction cycle.
  4. Carboplatin + Pemetrexed: Carboplatin AUC 5 and pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for 4 cycles.
  Radiation: Either standard 3DCRT or IMRT was delivered using EBRT of 5 fractions per week for ~6 weeks (± 3 days).
- Total: Total of all reporting groups
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT | Total
Number analyzed (Participants) | 219 | 109 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.96) | 62.4 (9.50) | 62.6 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 29 | 82
  Male | 166 | 80 | 246
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 141 | 62 | 203
  Black or African American | 2 | 0 | 2
  Asian | 65 | 39 | 104
  American Indian or Alaska Native | 7 | 7 | 14
  Other | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 21 | 54
  Not Hispanic or Latino | 186 | 88 | 274

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The PFS per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) using blinded independent central review (BICR) assessments was defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anti-cancer therapy prior to progression. The PD was defined as at least a 20% increase in the sum of diameters of target lesions. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at screening, 16 weeks ±1 week after randomization, then every 8 weeks ±1 week up to 48 weeks, and then every 12 weeks ±1 week thereafter until confirmed PD. Assessed up to the DCO date (a maximum of approximately 1988 days).
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
months | 13.8 [9.5 to 16.9] | 9.4 [7.5 to 16.6]
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; The hazard ratio (HR) and confidence intervals (CIs) were calculated using a stratified Cox proportional hazards model, adjusting for age [< 65 versus (vs.) >= 65 years] and stage (IIIA vs. IIIB/C), with treatment as the only covariate and ties handled by Efron approach; Test type: Superiority; p = 0.247, Log Rank; The analysis was performed using the stratified log-rank test, adjusting for age (< 65 vs. >= 65 years) and stage (IIIA vs. IIIB/C); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.647 to 1.123]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR per RECIST 1.1 using BICR was defined as the percentage of participants with a confirmed response of complete response (CR) or partial response (PR) based on all participants in the FAS. The CR was defined as disappearance of all target lesions since baseline. The PR was defined as at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: as for outcome 1
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
percentage of participants | 60.7 [53.9 to 67.2] | 60.6 [50.7 to 69.8]
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; Test type: Superiority; p = 0.976, Cochran-Mantel-Haenszel; The analysis was performed using a Cochran-Mantel-Haenszel (CMH) test, stratified by age (< 65 vs. >= 65 years) and stage (IIIA vs. IIIB/C); Difference in percentages = 0.2, 99.50% CI 2-sided [-15.2 to 16.3] — The CIs for difference in percentages were estimated using Miettinen and Nurminen's method

3. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of randomization until death due to any cause regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: From screening until confirmed PD, assessed up to the DCO date (a maximum of approximately 1988 days).
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
months | 36.4 [26.2 to 45.6] | 29.5 [23.2 to 45.1]
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; Test type: Superiority — The HR and CIs were calculated using a stratified Cox proportional hazards model, adjusting for age (< 65 vs. >= 65 years) and stage (IIIA vs. IIIB/C), with treatment as the only covariate and ties handled by Efron approach; p = 0.823, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.778 to 1.386]

4. Secondary Outcome: Percentage of Participants Alive at 24 Months From Randomization (OS24)
Description: The OS24 was defined as the Kaplan-Meier estimate of OS at 24 months. Median OS24 was calculated using the Kaplan-Meier technique.
Time Frame: Month 24
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
percentage of participants | 58.4 [51.6 to 64.7] | 59.5 [49.6 to 68.2]
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; Test type: Superiority — For the comparison between treatments, the Kaplan-Meier estimator of survival at 24 months for each treatment was used to obtain the HR and the test is based on the method described in Klein 2007. To account for the stratification factors, the estimates and test statistics in each strata were combined by weighting inversely proportionately according to each within stratum variance; p = 0.847, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.716 to 1.502]

5. Secondary Outcome: Complete Response Rate (CRR)
Description: The CRR per RECIST 1.1 using BICR was defined as the percentage of participants with a confirmed response of CR. The CR was defined as disappearance of all target lesions since baseline.
Time Frame: as for outcome 1
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
percentage of participants | 1.8 [0.5 to 4.6] | 1.8 [0.2 to 6.5]
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; Test type: Superiority — The analysis was performed using a CMH test, stratified by age (< 65 vs. >= 65 years) and stage (IIIA vs. IIIB/C); Difference in percentages = 0.0, 95% CI 2-sided [-4.8 to 3.0] — The CIs for difference in percentages was calculated using Miettinen and Nurminen's method

6. Secondary Outcome: Duration of Response (DoR)
Description: The DoR per RECIST 1.1 using BICR was defined as the time from the date of first documented response (which was subsequently confirmed) until the first date of documented progression or death in the absence of PD. The CR was defined as disappearance of all target lesions since baseline. The PR was defined as at least a 30% decrease in the sum of the diameters of target lesions. The DoR was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: The FAS included all randomized participants. Only participants with objective response are analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 133 | 66
months | 30.7 [8.8 to NA] — Upper limit of inter-quartile range could not be calculated as it was not reached as there were an insufficient number of participants with events. | 18.6 [7.4 to 56.5]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR at 24 weeks per RECIST 1.1 using BICR was defined as the percentage of participants who had a best objective response of CR or PR in the first 25 weeks (to allow for late assessment within the assessment window) or who had stable disease for >= 23 weeks after randomization (to allow for an early assessment within the ± 1 week assessment window).
Time Frame: Week 24
Population: The FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
percentage of participants | 65.8 | 65.1

8. Secondary Outcome: Time to Death or Distant Metastasis (TTDM)
Description: The TTDM per RECIST 1.1 using BICR was defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis. Distant metastasis was defined as any new lesion that was outside the radiation field according to RECIST 1.1 or proven by biopsy.
Time Frame: as for outcome 1
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
months | 51.0 [25.0 to NA] — Upper limit of inter-quartile range could not be calculated as it was not reached as there were an insufficient number of participants with events. | 46.3 [16.6 to NA] — Upper limit of inter-quartile range could not be calculated as it was not reached as there were an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.790, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.649 to 1.413]

9. Secondary Outcome: Time From Randomization to Second Progression (PFS2)
Description: The PFS2 was defined as the time from the date of randomization to the earliest of the progression event (subsequent to that used for the primary variable PFS per Investigator assessment) or death. The date of the second progression was recorded by the Investigator and defined according to local standard clinical practice and could have involved any of objective radiological, symptomatic progression, or death. Median PFS2 was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 109
months | 27.8 [21.8 to 35.8] | 22.0 [16.2 to 28.0]
Statistical Analysis 1: Comparison: Durvalumab + SoC CRT vs Placebo + SoC CRT; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.132, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.614 to 1.071]

10. Secondary Outcome: Serum Concentration of Durvalumab
Description: Blood samples were collected to determine the concentration of durvalumab.
Time Frame: End of infusion on Week 0, pre-infusion on Weeks 4 and 12, and Month 3 follow-up
Population: The Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of durvalumab or matching placebo per protocol, for whom any post-dose data were available and did not violate or deviate from the protocol in ways that would significantly affect the PK analyses. Only participants analyzed at specific timepoint are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Arm/Group | Durvalumab + SoC CRT
Number analyzed (Participants) | 190
microgram per milliliter
  Week 0: End of infusion | 452.21 (78.94)
  Week 4: Pre-infusion: number analyzed (Participants) | 179
  Week 4: Pre-infusion | 82.02 (80.85)
  Week 12: Pre-infusion: number analyzed (Participants) | 132
  Week 12: Pre-infusion | 123.39 (163.20)
  Month 3 Follow-up: number analyzed (Participants) | 39
  Month 3 Follow-up | 15.79 (243.41)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: Blood samples were collected to determine the presence of ADAs and ADA-neutralizing antibodies (nAb) for durvalumab using validated assays. ADA prevalence was defined as the number of participants with positive ADA result at any time, baseline or post-baseline. ADA incidence was defined as either treatment-induced (post-baseline ADA positive only) or treatment-boosted ADA (baseline positive ADA titer that was boosted to >= 4-fold during the study period). Treatment-induced ADA was defined as ADA positive only post-baseline and not detected at baseline. Persistently positive was defined as having at least 2 post-baseline ADA positive assessments with at least 16 weeks between the first and last positive assessment, or ADA positive at the last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment without fulfilling the conditions for persistently positive.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2 and 4
Population: The ADA analysis set included all participants who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + SoC CRT
Number analyzed (Participants) | 199
Participants
  ADA positive at any visit (ADA prevalence) | 20
  Treatment-emergent ADA positive (ADA incidence) | 8
  ADA positive at both baseline and post-baseline | 2
  Treatment-induced ADA | 8
  ADA positive at baseline only | 10
  Treatment-boosted ADA | 0
  Persistent positive | 6
  Transient positive | 4
  nAb positive at any visit | 1

12. Secondary Outcome: Change From Baseline in Disease-Related Symptoms as Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC QLQ) at Average Over 12 Months
Description: Patient reported outcomes for 5 disease related symptoms was assessed using the EORTC QLQ-Core 30 (C30) items questionnaire (fatigue and appetite loss) and the EORTC QLQ-Lung Cancer module 13 (LC13) (dysponea, cough and chest pain). An outcome variable consisting of a total score from 0 to 100 was derived for each of the symptom scales/symptom items, the functional scales, and the global health status scale with higher scores on the global health status/quality of life (QoL) and functioning scales representing better health status/function, but higher scores on symptom scales/items representing greater symptom severity. An improvement in symptoms were indicated by a negative change in score from baseline. A positive change in score from baseline indicated a deterioration of symptoms. A minimum clinically meaningful change was defined as a change from baseline of >=10.
Time Frame: At screening, 2, 4, 6, 8, 12, 16, and 20 weeks after randomization, then every 8 weeks ±1 week up to 52 weeks, and then every 12 weeks ±1 week thereafter until PFS2. Assessed up to 12 months.
Population: The FAS included all randomized participants. Only participants analyzed at baseline through Month 12 are reported.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 196 | 95
units on a scale
  EORTC QLQ-C30: Global health status/QoL | -0.5 [-2.3 to 1.4] | 0.2 [-2.4 to 2.8]
  EORTC QLQ-C30: Physical functioning | -1.4 [-3.0 to 0.2] | -0.8 [-3.1 to 1.4]
  EORTC QLQ-C30: Fatigue symptoms | 1.3 [-0.9 to 3.4] | 0.3 [-2.8 to 3.3]
  EORTC QLQ-C30: Appetite loss symptoms | 3.0 [0.9 to 5.2] | 0.3 [-2.7 to 3.3]
  EORTC QLQ-LC13: Dyspnoea symptoms | 1.1 [-1.0 to 3.1] | -1.3 [-4.2 to 1.6]
  EORTC QLQ-LC13: Cough symptoms | -6.1 [-8.6 to -3.6] | -6.5 [-10.0 to -2.9]
  EORTC QLQ-LC13: Pain in chest symptoms | -1.9 [-4.2 to 0.4] | -0.8 [-3.9 to 2.4]

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is the development of any untoward medical occurrence in a participant or clinical study participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A SAE is an AE occurring during any study phase, that fulfils 1 or more of the following criteria: death, life-threatening, in-participant hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital abnormality or birth defect, and an important medical event that may jeopardize the participant or may require medical treatment to prevent 1 of the outcomes listed above. AEs leading to discontinuation of study treatment were those with action taken was 'Drug Permanently Discontinued' for any study treatment.
Time Frame: From time of signature of informed consent up to 90 days after last dose of study treatment or up to the date of initiation of the first subsequent therapy, whichever occurs first, approximately 1988 days.
Population: The Safety analysis set included all participants who received at least 1 dose of randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
Number analyzed (Participants) | 219 | 108
percentage of participants
  Any AE | 98.6 | 100.0
  Any SAE | 47.0 | 51.9
  Any AE leading to discontinuation of treatment | 34.7 | 19.4
  Any immune-mediated AE | 48.9 | 28.7

ADVERSE EVENTS:
Time Frame: From time of signature of informed consent up to 90 days after last dose of study treatment or up to the date of initiation of the first subsequent therapy, whichever occurs first, approximately 1988 days.
Description: The Safety analysis set included all participants who received at least 1 dose of randomized treatment. All-cause mortality was determined for participants in FAS.
Arm/Group | Durvalumab + SoC CRT | Placebo + SoC CRT
All-Cause Mortality (participants affected / at risk) | 142/219 | 69/109
Serious Adverse Events (participants affected / at risk) | 103/219 | 56/108
Other Adverse Events (participants affected / at risk) | 209/219 | 106/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + SoC CRT (N=219) | Placebo + SoC CRT (N=108)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 5 (5)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 29 (37) | 11 (13)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 4 (4)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 1 (1)
Septic coagulopathy (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (4)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + SoC CRT (N=219) | Placebo + SoC CRT (N=108)
Nausea (Gastrointestinal disorders) | 55 (71) | 26 (30)
Odynophagia (Gastrointestinal disorders) | 14 (14) | 6 (7)
Oesophagitis (Gastrointestinal disorders) | 20 (20) | 8 (8)
Lymphopenia (Blood and lymphatic system disorders) | 29 (50) | 18 (27)
Vomiting (Gastrointestinal disorders) | 28 (32) | 7 (9)
Asthenia (General disorders) | 30 (35) | 8 (11)
Fatigue (General disorders) | 36 (41) | 12 (13)
Pyrexia (General disorders) | 29 (38) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 59 (96) | 28 (33)
Bronchitis (Infections and infestations) | 10 (10) | 7 (7)
COVID-19 (Infections and infestations) | 13 (13) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 44 (56) | 19 (21)
Influenza (Infections and infestations) | 13 (15) | 3 (4)
Pneumonia (Infections and infestations) | 21 (22) | 15 (17)
Upper respiratory tract infection (Infections and infestations) | 13 (19) | 8 (10)
Urinary tract infection (Infections and infestations) | 16 (23) | 5 (6)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 38 (39) | 18 (18)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 33 (34) | 17 (18)
Radiation skin injury (Injury, poisoning and procedural complications) | 26 (26) | 11 (11)
Amylase increased (Investigations) | 18 (24) | 11 (16)
Blood creatinine increased (Investigations) | 10 (13) | 7 (10)
Lymphocyte count decreased (Investigations) | 10 (13) | 6 (7)
Neutrophil count decreased (Investigations) | 24 (35) | 8 (12)
Platelet count decreased (Investigations) | 17 (20) | 11 (14)
Anaemia (Blood and lymphatic system disorders) | 90 (105) | 40 (52)
Weight decreased (Investigations) | 24 (26) | 13 (15)
White blood cell count decreased (Investigations) | 18 (20) | 11 (14)
Decreased appetite (Metabolism and nutrition disorders) | 46 (51) | 21 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (33) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (25) | 14 (14)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 5 (7)
Dizziness (Nervous system disorders) | 11 (11) | 5 (11)
Headache (Nervous system disorders) | 18 (20) | 5 (5)
Insomnia (Psychiatric disorders) | 26 (30) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (55) | 18 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 8 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 8 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (16) | 13 (13)
Hyperthyroidism (Endocrine disorders) | 27 (28) | 5 (5)
Hypothyroidism (Endocrine disorders) | 36 (36) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (26) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 18 (20) | 9 (9)
Hypertension (Vascular disorders) | 18 (20) | 13 (15)
Abdominal pain upper (Gastrointestinal disorders) | 13 (15) | 5 (5)
Constipation (Gastrointestinal disorders) | 35 (43) | 31 (34)
Diarrhoea (Gastrointestinal disorders) | 30 (46) | 10 (18)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 12 (12)
Dysphagia (Gastrointestinal disorders) | 29 (29) | 9 (10)
Leukopenia (Blood and lymphatic system disorders) | 48 (80) | 19 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03519971/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03519971/SAP_002.pdf